CLINICAL TRIAL: NCT05598593
Title: Modified TBF Regimen as Conditioning Regimen Prior to Allogeneic Hematopoietic Cell Transplantation for T Cell Acute Lymphoblastic Leukemia/Lymphoblastic Lymphoma：Phase II Study
Brief Title: Modified TBF Regimen as Conditioning Regimen Prior to Allo-HSCT for T-ALL/LBL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZJU-HSCT-MTBF
Record Dates: First submitted 2022-10-26; First posted 2022-10-28 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Cytarabine+Thiotepa + Fludarabine + Busulfan; T Cell Acute Lymphoblastic Leukemia/Lymphoblastic Lymphoma
Keywords: allogeneic hematopoietic stem cell transplantation; T cell Acute Lymphoblastic Leukemia/Lymphoblastic lymphoma; thiotepa
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Busulfan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Modified TBF Conditioning Regimen (Experimental): thiotepa 5mg/kg/d d-9 to d-8, cytarabine 0-4.0 g/m2/d d-7 to d-6(adjusted according to patients' age and HCT-CI index), fludarabine 30mg/m2/d d-7 to d-3, busulfan 3.2mg/m2/d d-5 to d-3
  Interventions: Drug: cytarabine+thiotepa+ fludarabine + busulfan

INTERVENTIONS:
Drug: cytarabine+thiotepa+ fludarabine + busulfan — cytarabine+thiotepa+ fludarabine + busulfan intravenous injection

SUMMARY:
T cell acute lymphoblastic leukemia (T-ALL)/Lymphoblastic lymphoma (LBL) is a hematological malignancy caused by malignant transformation and clonal expansion of T-lineage precursor cells. The long-term cure rate of pediatric patients with T-ALL/LBL reaches 90%, but long-term survival of adult patients is less than 60%. Moreover, patients with high-risk factors such as PTEN/NRAS gene mutation, early T cell precursor (ETP) phenotype or positive minimal residual disease (MRD) have high rates of chemoresistance and dismal outcome. Allogeneic hematopoietic stem cell transplantation (allo-HSCT) can significantly improve the prognosis of high-risk T-ALL/LBL. Total body irradiation (TBI)-based conditioning chemotherapy regimen is the preferred regimen for allo-HSCT in children and young adults with ALL because of lower relapse rates and satisfactory survival. Different from children, the non-relapse-related mortality (NRM) after TBI-based preconditioning in adults (especially those >35 years old) was reported as high as 38%. In addition, serious sequelae after TBI seriously affect the quality of life and non-radiation conditioning chemotherapy regimens are urgently needed for T-ALL/LBL. The reported recurrence rates after BUCY (busulfan + cyclophosphamide) conditioning regimen for T-ALL as 41.2%. -56.7% and long-term survival was only 30-50%. Thiotepa is an ethyleneimine alkylating agent with anti-tumor effects and immunosuppressive effects, thus is widely used in conditioning regimen before HSCT. Retrospective paired analysis from EBMT indicated conditioning regimen thiotepa achieved similar relapse rates, long-term survival and faster granulocyte and platelet engraftment than TBI regimen. A recent retrospective study of childhood ALL from Turkey also reported that the TBF(thiotepa + fludarabine + busulfan) regimen had a recurrence rate of only 11.9% , a non-relapse mortality rate of 14.0% and a long-term survival of 79.1%. Data from a large retrospective paired study suggested TBF regimen can significantly reduce the relapse rate of acute myeloid leukemia after the first remission (HR=0.4, CI 0.2-0.7, P = .02) without increasing treatment related deaths compared with the traditional BUCY regimen. Based on these data, we modified the TBF regimen with additional cytarabine for allo-HSCT in T-ALL/LBL with expection to reduced disease relapse and improved long-term survival.

ELIGIBILITY:
Inclusion Criteria:

1. Age younger than 65 years
2. Patients diagnosed with T cell acute lymphoblastic leukemia/lymphoma , T-ALL/LBL according to WHO diagnostic criteria.
3. Patients who have donors and plane to accept allogeneic hematopoietic stem cell transplantation treatment.
4. ECOG body status score 0-2.
5. Good organ function level: ANC (neutrophil absolute value >=1.0x10^9/ L; PLT >=30x10^9/L; HB >=80g/L; Tibil <=1.5 ULN; ALT / AST <=2.5 ULN; bun / Cr <=1.5 ULN; LVEF >=50%).
6. Patients who voluntarily participate in the clinical trial, understand the research procedure and can sign the informed consent in writing.

Exclusion Criteria:

1. Patients who with severe cardiac insufficiency, cardiac ejection fraction EF is less than 60%; or severe arrhythmia, the investigator can not tolerate conditioning chemotherapy;
2. In patients with severe pulmonary insufficiency (obstructive and / or restrictive ventilation disorders), the researchers evaluated the patients who could not tolerate conditioning chemotherapy;
3. Patients with severe liver function impairment and liver function indexes (alt, TBIL) more than 3 ULN were evaluated as intolerant of conditioning chemotherapy;
4. In patients with severe renal insufficiency, the renal function index (CR) is more than 2 times of the upper limit of the normal value (ULN), or the 24-hour creatinine clearance rate (CR) is less than 50ml / min, the researchers evaluated that they could not tolerate conditioning chemotherapy;
5. In patients with severe active infection, the researchers evaluated that they could not tolerate conditioning chemotherapy;
6. Patients who had allergic reactions or serious adverse reactions in the previous use of pretreatment related drugs could not be included in the study.
7. Other reasons why the researchers could not be selected.

Ages: 4 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-10-23 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | 2 year
  2-year DFS

SECONDARY OUTCOMES:
incidence of toxic reaction | 2 year
  2-year incidence of toxic reaction
overall survival | 2 year
  2-year OS
umulative incidence of relapse | 2 year
  2-year incidence of relapse
ncidence of acute and or chronic graft verus host disease | 2 year
  2-year incidence of cGVHD

CONTACTS AND LOCATIONS:
Overall Officials: Yi Luo, M.D., Principal Investigator — First Affilaated Hospital of Medical School of Zhejiang University
Locations (1):
- The First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No